CLINICAL TRIAL: NCT05465434
Title: Study to Evaluate the Possible Antifibrotic Effect of Zinc Sulphate in Chronic HCV Patient Receiving Direct Acting Anti-viral Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dina Samir Ahmed Attalla, Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Clinical hepatology
Record Dates: First submitted 2022-07-13; First posted 2022-07-19 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 2 (Active Comparator): 25 patients will receive 50mg Zinc Sulphate plus the standard direct acting anti-viral therapy for 3 months.
  Interventions: Drug: Zinc Supplement
- Group 1 (No Intervention): 25 patients will receive their standard direct acting anti-viral therapy for 3 months

INTERVENTIONS:
Drug: Zinc Supplement — Zinc sulphate 50 mg
  Arms: Group 2

SUMMARY:
This study aims to evaluate the possible antifibrotic effect of zinc sulphate in chronic HCV patient receiving direct acting anti-viral therapy

DETAILED DESCRIPTION:
Chronic infection with hepatitis C virus (HCV) is a leading cause of liver-related morbidity and mortality worldwide and predisposes to liver fibrosis and end-stage liver complications. Liver fibrosis is the excessive accumulation of extracellular matrix proteins, including collagen, and is considered as a wound healing response to chronic liver injury.

Removal or elimination of the causative agent such as control or cure of viral infection has shown that liver fibrosis is reversible. Thus, there is a huge unmet medical need for anti-fibrotic therapies to prevent liver disease progression and Hepatocellular Carcinoma (HCC) development. However, while many anti-fibrotic candidate agents have shown robust effects in experimental animal models, but uptill now, no approved therapy exists for liver fibrosis.

The once-daily oral combination of Daclatasvir 60 mg and Sofosbuvir 400 mg once daily, for the treatment of non-cirrhotic naïve patients with chronic hepatitis C virus genotype 4 infection for 12 weeks, is effective and well tolerated in these patients.

Zinc, an essential trace element, is involved in the enzymatic activities and structural maintenance of numerous enzymes and proteins, and it has various physiological roles in the body. Specifically, zinc works as a growth factor and exerts immunomodulatory , antioxidant, anti-apoptotic and anti-inflammatory effects.

Zinc deficiency is prevalent in cirrhosis patients, whereas nitrogen metabolic disorders, particularly hypoalbuminemia, can be an indicator of zinc deficiency.

Zinc supplementation therapy has a great benefit in the management of chronic liver disease and seems to improve liver pathology and reduce the incidence of liver fibrosis and HCC.

It has been found that zinc supplementation inhibited liver inflammation and fibrosis in bile duct ligation (BDL) mice through selective suppression of M1 macrophages.

Therefore, oral zinc supplementation is recommended as a means of suppressing HCC development in patients who have achieved sustained virological response (SVR) after direct acting antiviral therapies (DAAs) treatment . Zinc is a powerful supplement not only to increase SVR in non-responders but also to improve hepatic functions and fibrosis.

Fibronectin (FN), which is produced by hepatic stellate cells (HSCs), is a multifunctional glycoprotein and extracellular matrix (ECM) component that is present in the cell membrane and cytoplasm and associated with cell cycle progression, participates in cell adhesion and proliferation, and has an important role in fibrotic progression, excessive FN deposition occurs prior to collagen deposition.

Fibronectin expression was gradually increased in response to TGFβstimulation of HSCs, It is a good noninvasive marker for the assessment of liver fibrosis in patients with chronic HCV.

Transforming growth factor (TGF)-β is a master profibrogenic cytokine and a promising target to treat fibrosis.

Hyaluronic acid is a chief component of the extracellular matrix (ECM) of connective tissues and plays the main structural role in the formation of ECM. The most important organ involved in the synthesis of hyaluronic acid is the liver and the results of clinical studies have shown its high diagnostic sensitivity in the pathological processes of the liver.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with fibrosis stage (F1&F2) post chronic HCV infection.

  * Age > 18 and < 65 years.

Exclusion Criteria:

* Patients with prior history of liver transplantation.
* Patients with prior history of hepatocellular carcinoma.
* Patients coinfected with HIV or HBV.
* Patients with any malignancies.
* Pregnant and lactating women.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Abdominal Ultrasonography | 3 months
  Assessment the change in the degree of liver fibrosis post treatment and compare their results before and post treatment
Serum fibronectin level | 3 months
  Fibronectin (FN), which is produced by hepatic stellate cells (HSCs), participates in cell adhesion and proliferation, and has an important role in fibrotic progression, excessive FN deposition occurs prior to collagen deposition
Serum transforming growth factor - beta 1 (TGF- β1) level | 3 months
  Transforming growth factor (TGF)-β is a good noninvasive marker for the assessment of liver fibrosis in patients with chronic HCV and also considered as a master profibrogenic cytokine and a promising target to treat fibrosis (15)
Fibrosis-4 (FIB-4) Score | 3 months
  The Fibrosis 4 score is a non-invasive scoring system based on several laboratory tests (AST/ALT/Platelets) that help to non-invasively estimate the amount of scarring in the liver. This score has been studied in liver disease due to Hepatitis C and Non-alcoholic steatohepatitis (NASH)
  FIB-4 = (Age (years)XAST Level (U/L))/(Platelet Count (〖10〗^9/L) X √(ALT (U/L)))
  FIB-4>3.25 confirms the presence of advanced fibrosis (F4)
  FIB-4<1.45 exclude the presence of advanced fibrosis (F3-F4)
  Values between 1.45 and 3.25 did not fully discriminate fibrosis and would need an additional method to predict liver fibrosis
AST to Platelet Ratio Index (APRI) score | 3 months
  The APRI model was developed as a simple, easily calculated method to predict significant, severe fibrosis (or cirrhosis) and has been tested in persons with HCV mono-infection and those with HCV and HIV Co-infection
  APRI = (AST Level /AST (Upper Limit of Normal))/(Platelet Count (〖10〗^9/L) )X100
  If the score is less than or equal to 0.5, the liver is either completely free of fibrosis (F0), or has a tiny bit of scarring (F1 or F2 by METAVIR Score).
  If the score is 1.5 or greater, the liver has scarring and likely some cirrhosis (F3 or F4 by METAVIR Score)
Serum hyaluronic acid level | 3 months
  Hyaluronic acid is a chief component of the extracellular matrix (ECM) of connective tissues and The most important organ involved in the synthesis of hyaluronic acid is the liver

CONTACTS AND LOCATIONS:
Locations (1):
- National Liver Institute, Shibīn al Kawm, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Haggar SM, Attalla DS, Elhelbawy M, El-Afify DR. A randomized clinical study to evaluate the possible antifibrotic effect of zinc sulfate in chronic HCV patient receiving direct-acting anti-viral therapy. Inflammopharmacology. 2025 Jan;33(1):329-339. doi: 10.1007/s10787-024-01628-3. Epub 2025 Jan 9. PMID 39789197
- See also: Chronic hepatitis C and liver fibrosis , Clinical studies with CHC patients demonstrated that non-invasive methods are in most cases accurate for diagnosis and for monitoring liver disease complications. Moreover, they have a high prognostic value — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4145747/
- See also: Liver Fibrosis: Mechanistic Concepts and Therapeutic Perspectives , ummarize cellular drivers and molecular mechanisms of fibrogenesis in chronic liver diseases and discuss their impact for the development of urgently needed anti-fibrotic therapies. — https://pubmed.ncbi.nlm.nih.gov/32260126/
- See also: Sustained virological response in patients with HCV treated with daclatasvir plus sofosbuvir, with or without ribavirin — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7747789/
- See also: Ledipasvir/Sofosbuvir versus Daclatasvir/Sofosbuvir for the Treatment of Chronic Hepatitis C Genotype 4 Patients — https://pubmed.ncbi.nlm.nih.gov/31573893/
- See also: Associations between Zinc Deficiency and Metabolic Abnormalities in Patients with Chronic Liver Disease — https://pubmed.ncbi.nlm.nih.gov/29342898/
- See also: Zinc and protein metabolism in chronic liver diseases — https://pubmed.ncbi.nlm.nih.gov/31891865/
- See also: Zinc deficiency as an independent prognostic factor for patients with early hepatocellular carcinoma due to hepatitis virus — https://pubmed.ncbi.nlm.nih.gov/31729124/
- See also: Long-Term Zinc Supplementation Improves Liver Function and Decreases the Risk of Developing Hepatocellular Carcinoma — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6316561/
- See also: Long-Term Zinc Supplementation Improves Liver Function and Decreases the Risk of Developing Hepatocellular Carcinoma — https://pubmed.ncbi.nlm.nih.gov/34614431/
- See also: Selective suppression of M1 macrophages is involved in zinc inhibition of liver fibrosis in mice — https://pubmed.ncbi.nlm.nih.gov/34119631/
- See also: Oral Zinc Supplementation Decreases the Risk of HCC Development in Patients With HCV Eradicated by DAA — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8631098/
- See also: IL28B rs12979860 polymorphism and zinc supplementation affect treatment outcome and liver fibrosis after direct-acting antiviral hepatitis C therapy — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8501168/
- See also: Zinc Administration and Improved Serum Markers of Hepatic Fibrosis in Patients with Autoimmune Hepatitis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8199625/
- See also: Value of serum fibronectin for assessment of liver fibrosis in chronic hepatitis C virus patients — https://ejim.springeropen.com/articles/10.4103/ejim.ejim_46_19
- See also: TGF-β in Hepatic Stellate Cell Activation and Liver Fibrogenesis — https://pubmed.ncbi.nlm.nih.gov/31718044/
- See also: Hyaluronic acid as a potential marker for assessment of fibrosis regression after direct acting antiviral drugs in chronic hepatitis C patients — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8527342/
- See also: Advances in non-invasive assessment of hepatic fibrosis — https://pubmed.ncbi.nlm.nih.gov/32066623/